CLINICAL TRIAL: NCT06211205
Title: Effectiveness of a Customized 3D Printed Nostril Retainer Combined With Taping Vs. Taping Only on Enhancing the Nasolabial Esthetics and Maxillary Arch Dimensions in Infants With Unilateral Complete Cleft Lip and Palate: A Randomized Clinical Trial.
Brief Title: Effectiveness of a Customized 3D Printed Nostril Retainer Combined With Taping Vs.Taping Only on Enhancing the Nasolabial Esthetics and Maxillary Arch Dimensions in Infants With Unilateral Complete Cleft Lip and Palate.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hana Adel Adawy, Hana Adawy, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCT26091993123
Record Dates: First submitted 2023-12-24; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Cleft Lip and Palate
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Customized nostril retainer combined with lip taping (Experimental)
  Interventions: Device: Customized 3D printed nostril retainer combined with lip taping
- Lip taping (Active Comparator)
  Interventions: Procedure: Lip taping

INTERVENTIONS:
Device: Customized 3D printed nostril retainer combined with lip taping — the infants will receive a customised nostril retainer appliance to enhance the nasal esthetics combined with lip tape to approximate the labial and alveolar segments
  Arms: Customized nostril retainer combined with lip taping
Procedure: Lip taping — the infants will receive lip tape to approximate the labial and alveolar segments
  Arms: Lip taping

SUMMARY:
Lip taping was proven as simple, handy technique of PSIO for alveolar molding yielding enhanced maxillary arch dimensions in UCCLP infants.

The approach behind this study is to combine this simple step with a digitally designed 3D printed customized nasal molding device to enhance the naslolabial esthetics and maxillary arch dimensions in infants with unilateral complete cleft lip and palate, employing full digital workflow.

ELIGIBILITY:
Inclusion Criteria:

1. Infants with age range from 1-30 days.
2. Unilateral complete cleft lip and palate
3. Medically free subjects.
4. Both males and females.

Exclusion Criteria:

1. Patients older than 30 days.
2. Syndromic patients with other defects in addition to cleft lip and palate.
3. Patients with bilateral cleft lip and palate.
4. Incomplete cleft lip.
5. Patient with previous surgical lip repair or adhesion.
6. Patients with previous presurgical infant orthopedic treatment.
7. Medically compromised patients.

Max Age: 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-01-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Nasolabial esthetics | 3 months
  Nasal basal width, Collumella Length, Defetcted Nostril width and height, Interlabial gap will be measured in mm at 2 time points to evaluate the effect of the intervention.
  This will be performed on a 3D scan for the infants and through calibrated photographs

SECONDARY OUTCOMES:
Maxillary arch changes | 3 months
  Interalveolar gap will be measured in mm through an intraoral scan for the infants at 2 time points

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthodontics, Faculty of Dentistry, Cairo university, Cairo, Egypt